CLINICAL TRIAL: NCT04694313
Title: Evaluation of Optical Pumping Magnetometer Sensors for MagnetoEncephaloGraphy Imaging
Acronym: OPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-43; 2020-A01830-39 (Other: ID-RCD)
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPM (Experimental): Two types of measurement will be compared (SQUID and OPM) with the reference that constitutes the in-depth recordings (Stereotactic-EEG or SEEG) used to precisely define the region of the brain to be resected in order to cure epileptic patients of their seizures.
  Interventions: Device: OPM

INTERVENTIONS:
Device: OPM — Simultaneous MEG SQUID + SEEG acquisition followed by a simultaneous MEG OPM + SEEG acquisition.

SUMMARY:
This research is a feasibility study on a new generation of brain magnetic activity sensor which should allow the development of this modality, until now limited by its cost to a few large university centers.

The measurement of magnetic activity allows the detection and localization of abnormal activities such as paroxysmal events occurring between seizures in patients with epilepsy as well as research into brain function. It is the only one, along with EEG and related techniques, to provide data related to the speed of the brain. MEG, by virtue of the properties of magnetic fields, has a greater potential than EEG for the detection and localization of the neuronal sources which cause it.

The MEG sensors used until now use Superconducting Quantum Interference Devices (SQUID) components that are extremely sensitive but require complex instrumentation and only operate under superconducting conditions, resulting in prohibitive maintenance and cost.

The alternative could come from a new magnetic activity sensor: the optical pumping magnetometers of the alkaline type.

This preliminary study proposes to compare SQUID sensors with MPO He4 sensors for their ability to detect abnormal activities recorded in epileptic patients. Measurements that cannot be recorded simultaneously Two types of measurement will be compared with the reference that constitutes in-depth recording (Stereotactic-EEG or SEEG) used to precisely define the region of the brain to be resected in order to cure epileptic patients of their seizures.

The expected results are a capacity of this type of sensors to detect epileptic activities equivalent to that of SQUIDs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Patient with drug-resistant focal epilepsy, undergoing SEEG exploration
* Healthy subject, devoid of central neurological pathology, major ((≥ 18 years)
* Patient or healthy subject capable of giving informed consent for the study

Exclusion Criteria:

* MEG "incompatible" healthy patients or volunteers.
* Wearers of prosthesis or pacemaker likely to generate artefacts interfering with the measurement. There is no danger to the subject, but the measurement itself may be impossible.
* Patients or healthy volunteers who cannot stand standing still for a few minutes.
* Pregnant or breastfeeding women
* Adults under guardianship or under legal protection
* People deprived of their liberty
* People who have not signed the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Signal to noise ratio visible on the sensors | Visit 0 at month 0
  Interictal peaks or oscillations in different frequency bands (gamma, ripples, fast ripples)

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Department of Epileptology and Cerebral Rhythmology, Hôpital La Timone, APHM, Marseille, France

IPD SHARING:
Plan to Share IPD: No